CLINICAL TRIAL: NCT00443157
Title: A Phase II, Open Label, Randomised, Single Centre Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Three or Four Doses of Meningococcal Serogroup B Outer Membrane Vesicle (OMV) Vaccine MENZBTM When Administered to Healthy Adults (University Students)
Brief Title: Meningococcal B Vaccination in University Students
Acronym: MNB3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Public Health England (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MNB3
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2007-09

CONDITIONS: Neisseria Meningitidis Serogroup B
Keywords: meningococcal B vaccine

INTERVENTIONS:
Biological: Meningococcal B Vaccine NZ

SUMMARY:
This study is the third in a series using the MenB vaccine from the National Institute of Public Health in Norway (NIPH). The vaccine was first made in response to a high incidence of disease using the 44/76 strain which was resopnsible for most of the disease there. The VEC did the first study, MNB1, using this vaccine. Since then the NIPH has formed a commercial partnership with Chiron Vaccines and has reformulated the vaccine using the NZ98/254 MenB strain for use in New Zealand.

The vaccine was first produced at NIPH facilties and it was this vaccine that was used in our second study, MNB2. The current study, MNB3, will use the NZ98/254 MenB vaccine but from Chiron facilities where production has been scaled up in order to provide enough doses for the national immunisation campaign that is ongoing in New Zealand.

ELIGIBILITY:
Inclusion Criteria:

* Informed written consent given for four immunisations (group 2 will receive 3 doses only) with MeNZB TM vaccine, as well as for eight blood draws to be taken as described in the patient information leaflet in appendix 2
* Healthy adults (university students) aged 18 up to 40 years on inclusion in the study

Exclusion Criteria:

On enrolment:

* Previous history of bacteriologically confirmed disease caused by N. meningitidis
* Prior receipt of any group B meningococcal vaccine
* have had household contact with and/or intimate exposure to an individual with culture or PCR proven N. meningitidis serogroup B within the previous 60 days
* have either received, or for whom there is intent to immunize with, any vaccines or investigational agents within 50 days prior to enrolment, through to 50 days following the last study vaccine administration, with the exception of influenza vaccines or post-exposure tetanus vaccination
* have a history of any anaphylactic shock, urticaria or other allergic reaction after previous vaccinations or hypersensitivity to any vaccine component
* have experienced significant acute or chronic infections requiring systemic antibiotic treatment within the past 14 days
* have any present or suspected serious acute or chronic disease such as: cardiac or autoimmune disease, insulin dependent diabetes or progressive neurological disease or severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease; leukaemia, lymphomas, neoplasm;
* have a known or suspected impairment of the immune function, or those receiving immunosuppressive therapy, or having received immunosuppressive therapy, including systemic steroids, or ACTH or inhaled steroids in dosages which are associated with hypothalamic-pituitary-adrenal axis suppression;
* have received blood, blood products or a parenteral immunoglobulin preparation in the past 12 weeks;
* have a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time;
* have a history of seizure disorder;
* have an inherited genetic anomaly (known cytogenic disorders) e.g., Down's syndrome;
* Language difficulty sufficient to preclude adequate comprehension of the information sheet, consent form or study nurse's explanation of the study;
* The possibility of pregnancy - a pregnancy test (urine) on the scheduled day of vaccination will be offered to any female wishing to participate in the study. A positive test will result in exclusion from the study. (Agreement from each female participants will be sought prior to vaccination that they will take adequate precautions to avoid pregnancy for the duration of the vaccination phase of the study until the final blood sample appointment following their final vaccination, i.e. until the week 63 - visit 8 - blood appointment);
* Current regimen of chronic prescription medications other than oral contraceptives, or current regular use of any over-the-counter concomitant medications including antipyretics and non-steroidal anti-inflammatory agents;
* Current participation in any other clinical trial (an undertaking will be sought from participants not to enrol in any other clinical trial for the duration of this study);
* They have any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives

Current (to be checked prior to each vaccination):

* Generalised acute systemic illness on the day of immunisation
* Sublingual temperature >38,5oC on the day of immunisation
* Development of any condition specified in the initial exclusion criteria cited above will constitute a criterion for exclusion from receiving subsequent vaccine doses.
* Any serious reaction related to the study vaccines, which in the opinion of the investigator should alter the course of subsequent study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2006-02; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
serum bactericidal antibody

SECONDARY OUTCOMES:
Serum antibody ELISA
Immunoblotting
Opsonophagocytosis assay

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MBBS FRCPath, Principal Investigator — Public Health England
Locations (1):
- University of Sheffield Medical School, Sheffield, United Kingdom